CLINICAL TRIAL: NCT00407680
Title: Intensive Medical Treatment for Nephropathy Caused by Type 2 Diabetes With Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kitasato University (Other)
Collaborators: Tokai University (Other); Yokohama City University Medical Center (Other); St. Marianna University School of Medicine (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8417
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2007-10

CONDITIONS: Type 2 Diabetes Mellitus; Hypertension
Keywords: Type 2 diabetes mellitus; Hypertension; Angiotensin II Receptor Blocker; Diabetic nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Diabetic Nephropathies | interventions — Fluvastatin

INTERVENTIONS:
Drug: Intensive therapy Valsartan,Fluvastatin

SUMMARY:
To observe the effect of intensive medical treatment for type 2 diabetic patients with hypertension: to discover whether or not intensive medical treatment improves proteinuria, and the difference between the clinical meaning of responder and non-responder (criteria: 50% reduced proteinuria continuing 6 months or more during the observation period.)

DETAILED DESCRIPTION:
It is reported that the risk of a cardiovascular event occurring is 1.78 times higher in patients with diabetic nephropathy (DN) than in patients without DN. It is also reported that angiotensin II receptor blockade (ARB) prevents the progression of DN in diabetic patients with early phase nephropathy beyond its blood pressure lowering effect. The guidelines by the Japanese Society of Hypertension 2004 recommended that it was necessary to control blood pressure (BP) below 130/80 mmHg in all diabetic patients. This has become the universal target BP for the prevention of cardiovascular events in hypertensive patients. On the study of intensive medical treatment [including angiotensin-converting enzyme inhibitor (ACEI)], it is reported that ACEI not only prevents the progression of DN in microalbuminuria but also decreases proteinuria <1 g/day in the nephrotic syndrome. Therefore, ACEI is thought to be effective for DN. However, it is not clear whether or not intensive medical treatment (including ACEI) improves nephropathy with proteinuria >1 g/day.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetic patients with hypertension, with all 5 of the criteria listed below:

1. Age 20 years and above
2. Blood pressure >125/75 mmHg
3. Urinary protein creatinine ratio 1g/g・cr or Urinary protein >1 g/day
4. Presence of diabetic retinopathy
5. Already performing dietary management

   * There were no limitations on serum creatinine.
   * BP was recorded 3 times while the patient was seated and averaged.
   * The subjects in this study were outpatients with written informed consent.

Exclusion Criteria:

1. Another definable renal disease other than DN
2. Collagenosis
3. Malignant hypertension with emergent treatment
4. Severe hypertension (diastolic BP >120 mmHg)
5. Severe chronic heart failure or acute myocardial infarction in the past 6 months
6. Atrial fibrillation or severe arrhythmia
7. Anamnesis of cerebrovascular disease with neuropathy
8. Anamnesis of anaphylaxis or chronic dermatopathy
9. Severe hepatic disease
10. Pregnancy
11. Anamnesis of anaphylaxis from angiotensin II receptor blocker
12. Patients are judged to be inapposite by the attending physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-10; Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Proteinuria
Serum Creatinine
e-GFR
Fasting Plasma Glucose
HbA1c

SECONDARY OUTCOMES:
Lipid profile
Blood pressure
Smoking
Progression of renal dysfunction
Urinary 8-OHdG,type 4 collagen,high molecular weight adiponectin
Serum angiotensinogen

CONTACTS AND LOCATIONS:
Overall Officials: Keiji Tanaka, MD,PhD, Study Chair — Kitasato University
Locations (1):
- Kitasato University, 1-15-1 Kitasato Sagamihara, Kanagawa, Japan